CLINICAL TRIAL: NCT06307600
Title: The Safety and Efficacy of RD06-03 CART Cell Injection in Patients With Relapsed or Refractory B-lymphoblastic Leukemia
Brief Title: The Safety and Efficacy of RD06-03 CART Cell Injection in Patients With R/R Acute B-lymphoblastic Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Chief Prof., Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-03-05
Record Dates: First submitted 2024-02-28; First posted 2024-03-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: B Lymphoblastic Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD06-03 cell infusion (Experimental): The enrolled patients will use 1 dose RD06-03 CART cell injection
  Interventions: Drug: RD06-03 cell injection

INTERVENTIONS:
Drug: RD06-03 cell injection — The patients in this intervention will use RD06-03 cell injection with 3 dose dose 1: 1×10^5 CAR+ T Cells/kg dose 2: 3×10^5 CAR+ T Cells/kg dose 3: 5×10^5 CAR+ T Cells/kg Dosage form: IV injection Frequency of administration：1 time
  Other Names: RD06-03

SUMMARY:
This study is designed to explore the safety and efficacy for patients with relapsed and/or refractory B-cell lymphoblastic leukemia.

DETAILED DESCRIPTION:
The study completes the enrollment of all evaluable subjects for DLT during the dose escalation phase, followed by DLT observation, and enters a efficacy exploration phase lasting up to 1 year. After safety conclusions are drawn for each group, investigators may choose to expand cases in the corresponding dose group based on treatment response, but the total number of cases should not exceed 12 (expanded cases are not subjected to DLT evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥3 and ≤70 years, gender and race unrestricted.
* Bone marrow examination confirms the diagnosis of acute B-cell lymphoblastic leukemia (B-ALL) and meets one of the following conditions:

Relapsed B-ALL: ① Relapse within 12 months after the first remission; or ② Relapse after salvage chemotherapy in first-line/multi-line treatment; or ③ Relapse after autologous or allogeneic hematopoietic stem cell transplantation; Refractory B-ALL: ① Failure to achieve complete remission after 2 cycles of standardized induction chemotherapy; or ② Failure to achieve complete remission after salvage chemotherapy in first-line/multi-line treatment;

* Ph+ALL subjects are eligible if they meet one of the following criteria: ① Relapse or refractory after receiving at least 2 tyrosine kinase inhibitors (TKIs) treatments; if accompanied by TKI-resistant mutations such as T315I/A, V299L, F317L/V/I/C, G250E, Y253H, E255K/V, F359V/C/I, subjects are not required to receive at least two TKI treatments; or ② Unable to tolerate TKI treatment; or ③ Contraindications to TKI treatment.
* The proportion of bone marrow blasts during the screening period is ≥5% (morphological).Expression of CD19 on bone marrow or peripheral blood tumor cells is detected during the screening period.
* Organ function and laboratory tests meet the following criteria:

Serum total bilirubin <2× upper limit of normal (ULN), serum ALT and AST both <3× ULN, serum creatinine <1.5× ULN; Coagulation function: International normalized ratio (INR) ≤1.5× ULN, or prothrombin time (PT) ≤1.5× ULN; Transthoracic echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%; Resting oxygen saturation (SpO2) ≥92% in ambient air; Estimated survival period of more than 3 months;

* ECOG score 0-2;
* Fertile women must agree to use highly effective contraception from at least 28 days before leukapheresis to 6 months after CAR-T cell infusion. Their partners, fertile men, must agree to use effective barrier contraception from the start of leukapheresis to 6 months after CAR-T cell infusion, and should not donate semen or sperm during the entire trial period.

Exclusion Criteria:

* Suffering from genetic syndromes such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndromes;
* History of allergy to any component of the cellular product;
* Presence of active central nervous system leukemia (CNSL) at screening;
* Patients with purely extramedullary relapse;
* Received allogeneic hematopoietic stem cell transplantation (HSCT) within 3 months before screening or experienced grade II to IV active graft-versus-host disease (GVHD) within 4 weeks before infusion;
* Significant cardiovascular dysfunction within 12 months before screening, including but not limited to: New York Heart Association (NYHA) class III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias.

Presence or suspicion of uncontrollable active infection requiring intravenous therapy (excluding simple urinary tract infections, bacterial pharyngitis);

* Subjects with a history of other primary cancers, excluding the following:

Non-melanoma skin cancers such as basal cell carcinoma that have been cured by resection; Cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ with disease-free survival ≥2 years after adequate treatment;

* Subjects with autoimmune diseases requiring treatment, immunodeficiency, or requiring immunosuppressive therapy;
* Received live attenuated vaccines within 4 weeks before screening, or planned to receive live attenuated vaccines during the study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 2 years
  DLT

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, phd, Principal Investigator — Anhui Provincial Hospital
Locations (2):
- China (2):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No